CLINICAL TRIAL: NCT01748448
Title: Vitamin D Supplementation in Cutaneous Malignant Melanoma Outcome
Acronym: ViDMe
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2012LRDVDCM; 2012-002125-30 (EudraCT Number)
Record Dates: First submitted 2012-12-05; First posted 2012-12-12 (Estimated); Results first posted 2025-02-17 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2023-03

CONDITIONS: Cutaneous Malignant Melanoma
Keywords: Cutaneous malignant melanoma; Vitamin D; Cholecalciferol
MeSH Terms: conditions — Melanoma, Cutaneous Malignant | interventions — Vitamin D; Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vitamin D (Active Comparator): Every month 100 000 units of Vitamin D in syringe oral dispenser is taken . Study duration is maximum 3,5 years or until relapse occurs
  Interventions: Drug: Vitamin D
- Placebo: Oil (Placebo Comparator): Every month 100 000 units of vitamin D in syringe Oral dispenser is taken. Study duration is maximum of 3.5 years or until relapse occurs
  Interventions: Drug: Placebo: Oil

INTERVENTIONS:
Drug: Vitamin D — * prospective interventional randomized double blind placebo controlled trail
  * clinical setting (tertiary university hospital)
  * investigator driven, no pharmaceutical sponsor
  * cutaneous malignant melanoma patients
  * add- on study (placebo or vitamin D) on top of optimal standard care
  * 1:1 inclusion ratio (placebo:Vitamin D)
  * randomisation after informed consent and screening
  Other Names: D-Cure; Cholecalciferol
  Arms: Vitamin D
Drug: Placebo: Oil
  Other Names: Placebo
  Arms: Placebo: Oil

SUMMARY:
To assess whether vitamin D supplementation after surgery of a first cutaneous malignant melanoma protects against relapse of the disease.

DETAILED DESCRIPTION:
To assess whether vitamin D supplementation, in the follow up period after diagnosis and surgery of a first cutaneous malignant melanoma, has a protective effect on relapse of cutaneous malignant melanoma and whether this protective effect correlates with vitamin D levels in serum and vitamin D receptor (VDR) immunoreactivity in the primary tumor.

ELIGIBILITY:
Inclusion Criteria:

1. Older than 18 years and younger than 80 years of age.
2. Histologically proven malignant melanoma, stage one B (IB) to three (III) Not participating in other clinical trial.
3. The only treatment for melanoma is surgical treatment.
4. Complete resection of melanoma.
5. Single primary invasive cutaneous melanoma
6. Signed ethical committee approved informed consent
7. Serum phosphate, serum calcium at the entry of the study within normal limits of laboratory reference

Exclusion criteria

1. Pregnant/lactating women or planning on becoming pregnant during the study
2. Known hypersensitivity to vitamin D or its components.
3. Pre-existing renal stone disease, chronic renal disease with glomerular filtration rate (eGFR) < 30 mL/min/1.73 m2 or renal dialysis.
4. Liver failure or chronic liver disease with liver enzymes > 2 fold upper limit of normal (ULN).
5. History of parathyroid disease or granulomatous disease (TBC and sarcoidosis)
6. History of malabsorption syndrome or any medical condition that might interfere with vitamin D absorption.
7. History of small intestine resection.
8. History of other malignancy within the last 5 years except for carcinoma in situ of the cervix or basal cell carcinoma or squamous cell carcinoma of the skin or in situ malignant melanoma.
9. Chronic alcohol abuse.
10. Medical or logistic problems likely to preclude completion of the study.
11. Taking medication that predisposes to hypercalcemia (digoxin, lithium, thiazide diuretics) or taking medication that would affect metabolism of vitamin D (anticonvulsants, corticosteroids, H2-receptor antagonists)
12. Intake of vitamin D supplements within 6 months prior to entry of the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 436 (Actual)
Dates: Start 2012-12 (Actual); Primary Completion 2022-07 (Actual); Study Completion 2022-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marjan Garmyn, MD, PhD, Principal Investigator — Universitaire Ziekenhuizen KU Leuven
Locations (4):
- Belgium (3):
  - Universitair Ziekenhuis Antwerpen, Dermatology, Edegem
  - UZLeuven Gasthuisberg, Leuven
  - Chef de Service du Service Universitaire de Dermatologie, Liège
- Dep. of Dermatology, Medical and Health Science Center University of Debrecen, Debrecen, Hungary

REFERENCES:
- [Background] De Smedt J, Van Kelst S, Boecxstaens V, Stas M, Bogaerts K, Vanderschueren D, Aura C, Vandenberghe K, Lambrechts D, Wolter P, Bechter O, Nikkels A, Strobbe T, Emri G, Marasigan V, Garmyn M. Vitamin D supplementation in cutaneous malignant melanoma outcome (ViDMe): a randomized controlled trial. BMC Cancer. 2017 Aug 23;17(1):562. doi: 10.1186/s12885-017-3538-4. PMID 28835228
- [Result] De Smedt J, Van Kelst S, Janssen L, Marasigan V, Boecxstaens V, Bogaerts K, Belmans A, Vanderschueren D, Vandenberghe K, Bechter O, Aura C, Lambrechts D, Strobbe T, Emri G, Nikkels A, Garmyn M. High-dose vitamin D supplementation does not improve outcome in a cutaneous melanoma population: results of a randomized double-blind placebo-controlled study (ViDMe trial). Br J Dermatol. 2024 Nov 18;191(6):886-896. doi: 10.1093/bjd/ljae257. PMID 38913652
- [Result] De Smedt J, Aura C, Van Kelst S, Janssen L, Marasigan V, Boecxstaens V, Stas M, Bogaerts K, Belmans A, Cleynen I, Vanderschueren D, Vandenberghe K, Bechter O, Nikkels A, Strobbe T, Emri G, Lambrechts D, Garmyn M. Clinical and genetic determinants of vitamin D receptor expression in cutaneous melanoma patients. Melanoma Res. 2024 Apr 1;34(2):125-133. doi: 10.1097/CMR.0000000000000929. Epub 2024 Feb 13. PMID 38348498
- [Result] De Smedt J, Van Kelst S, Janssen L, Marasigan V, Boecxstaens V, Stas M, Vanderschueren D, Guler I, Bogaerts K, Vandenberghe K, Bechter O, Billen J, Nikkels A, Strobbe T, Emri G, Lambrechts D, Garmyn M. Determinants of 25-hydroxyvitamin D Status in a Cutaneous Melanoma Population. Acta Derm Venereol. 2022 Apr 8;102:adv00692. doi: 10.2340/actadv.v102.262. PMID 35312026

RESULTS

PARTICIPANT FLOW:
Groups:
- Vitamin D: Every month 100 000 units of Vitamin D in syringe oral dispenser is taken . Study duration is maximum 3,5 years or until relapse occurs
  Vitamin D: - prospective interventional randomized double blind placebo controlled trail
  * clinical setting (tertiary university hospital)
  * investigator driven, no pharmaceutical sponsor
  * cutaneous malignant melanoma patients
  * add- on study (placebo or vitamin D) on top of optimal standard care
  * 1:1 inclusion ratio (placebo:Vitamin D)
  * randomisation after informed consent and screening
- Placebo: Oil: Every month 100 000 units of vitamin D in syringe Oral dispenser is taken. Study duration is maximum of 3.5 years or until relapse occurs
  Oil
Period: Treatment Period
Arm/Group | Vitamin D | Placebo: Oil
Started | 218 | 218
Completed | 216 | 217
Not Completed | 2 | 1
Not completed — Consent withdrawn by subject | 1 | 0
Not completed — Adverse Event | 1 | 0
Not completed — Personal | 0 | 1
Period: Follow-up Period
Arm/Group | Vitamin D | Placebo: Oil
Started | 216 | 217
Completed | 216 | 217
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vitamin D | Placebo: Oil | Total
Number analyzed (Participants) | 218 | 218 | 436
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 157 | 164 | 321
  >=65 years | 61 | 54 | 115
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 112 | 125 | 237
  Male | 106 | 93 | 199
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Education (highest level) [Count of Participants; unit: Participants]
  Primary | 9 | 8 | 17
  Secondary school | 75 | 68 | 143
  Vocational training | 43 | 40 | 83
  Vocational university | 62 | 59 | 121
  University graduated | 27 | 42 | 69
  Other | 1 | 1 | 2
  Unknown | 1 | 0 | 1
Current smoking [Count of Participants; unit: Participants]
  No | 99 | 76 | 175
  Yes | 33 | 37 | 70
  Never Smoked | 85 | 105 | 190
  Unknown | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Relapse Free Survival
Description: Disease free survival will be the primary endpoint of this phase III trial. Study duration for one patient is maximum 9 years and 7 months. Patients are supplemented with studymedication (Vitamin D or placebo) for maximum 3.5 years. This is the treatment period. After the treatment period (in which the patients take study medication, placebo or Vitamin D), there is the follow-up period, no more study medication is taken, the study is still double blind, and the patients are followed at the clinical department for relapse and/or death.
Time Frame: study duration maximum 9 years and 7 months or until relapse
Measure: Count of Participants; unit: Participants
Arm/Group | Vitamin D | Placebo: Oil
Number analyzed (Participants) | 218 | 218
Participants | 41 | 32
Statistical Analysis 1: Comparison: Vitamin D vs Placebo: Oil; Test type: Superiority; p = 0.324, Fisher Exact; Cox Proportional Hazard = 1.27, 95% CI 2-sided [0.79 to 2.03]

2. Secondary Outcome: Melanoma Subtype, as Assessed Clinically and Histologically
Description: Vitamin D levels at diagnosis will be correlated with melanoma subtype, as assessed clinically and histologically.
Time Frame: Time at diagnosis
Measure: Count of Participants; unit: Participants
Arm/Group | Vitamin D | Placebo: Oil
Number analyzed (Participants) | 217 | 218
Participants
  Nodular melanoma | 38 | 29
  Superficial spreading melanoma | 115 | 142
  Acrolentigineus melanoma | 8 | 6
  Lentigo maligna melanoma | 7 | 5
  Unknown | 22 | 21
  Other | 27 | 15

3. Secondary Outcome: Melanoma Site, as Clinically Recorded
Description: Vitamin D levels at diagnosis will be correlated with melanoma site, as clinically recorded.
Time Frame: Time at diagnosis
Measure: Count of Participants; unit: Participants
Arm/Group | Vitamin D | Placebo: Oil
Number analyzed (Participants) | 217 | 218
Participants
  Abdomen- chest | 18 | 26
  Arm - hand | 45 | 37
  Foot | 12 | 12
  Genitals | 1 | 2
  Head-neck | 31 | 27
  Leg | 55 | 61
  Back | 55 | 53

4. Secondary Outcome: 25(OH)D3 Serum Levels
Description: 25(OH)D3 serum levels will be recorded at diagnosis and at 6 months intervals up to final study visit.
Time Frame: study duration maximum 3.5 years (Treatment period) or until relapse
Population: The number of patients differs from baseline with the other time points for different reasons: patient was already End of study, no sample taken because of various reasons,...
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Vitamin D | Placebo: Oil
Number analyzed (Participants) | 214 | 218
ng/ml
  Baseline | 24 (9) | 23 (9)
  At Month 6: number analyzed (Participants) | 190 | 185
  At Month 6 | 43 (11) | 23 (9)
  At Month 12: number analyzed (Participants) | 148 | 143
  At Month 12 | 44 (11) | 24 (9)
  At Month 18: number analyzed (Participants) | 118 | 114
  At Month 18 | 44 (11) | 24 (11)
  At Month 24: number analyzed (Participants) | 82 | 87
  At Month 24 | 42 (11) | 24 (9)
  At Month 30: number analyzed (Participants) | 65 | 63
  At Month 30 | 44 (12) | 27 (8)
  At Month 36: number analyzed (Participants) | 39 | 45
  At Month 36 | 40 (12) | 25 (7)
  End of study (end of study medication): number analyzed (Participants) | 205 | 207
  End of study (end of study medication) | 43 (12) | 27 (9)

5. Secondary Outcome: Stage of Melanoma Patient
Description: Stage of melanoma patient at diagnosis according to the 8th American Joint Committee of Cancer (AJCC) Melanoma staging and classification.
  The eighth edition of the AJCC staging system is currently the most widely accepted and standardized approach to melanoma staging and classification at initial diagnosis. Melanoma staging is based on the American Joint Committee on Cancer (AJCC) staging system that uses three key pieces of information for assigning Tumor-Node-Metastasis (TNM) classifications. AJCC staging ifacilitates accurate risk stratification and is essential to guide patient treatment.
  The higher the stage, the more severe the melanoma.
Time Frame: Time at diagnosis
Measure: Count of Participants; unit: Participants
Arm/Group | Vitamin D | Placebo: Oil
Number analyzed (Participants) | 218 | 218
Participants
  IA | 24 | 26
  IB | 101 | 108
  IIA | 29 | 30
  IIB | 18 | 14
  IIC | 10 | 6
  IIIA | 14 | 10
  IIIB | 9 | 8
  IIIC | 10 | 14
  IIID | 0 | 1
  Unkown | 3 | 1

6. Other Pre Specified Outcome: Safety Endpoints:Incidence and Severity of Adverse Events
Description: Incidence and severity of adverse events will be recorded every 3 months up to final study visit (from the treatment period).
Time Frame: study duration maximum 3.5 years (Treatment period) or until relapse
Measure: Number; unit: Events
Arm/Group | Vitamin D | Placebo: Oil
Number analyzed (Participants) | 218 | 218
Events | 44 | 36

ADVERSE EVENTS:
Time Frame: In this study, the collection period for adverse events and serious Adverse events starts at the randomisation and ends when the patient completes the Treatment period of the study, serious and/or other adverse events were assessed up to 3.5 years. All-Cause Mortality was monitored for maximum 9 years and 7 months.
Description: The investigator will use the following terms te assess the severity of the adverse event: mild, moderate severe.
  The investigator will use the follwing causality terms to assess the relationship of teh adverse event or clinical efficacy to the use of the investigational medicinal product: reasonable causal relationship or not.
Arm/Group | Vitamin D | Placebo: Oil
All-Cause Mortality (participants affected / at risk) | 13/218 | 13/218
Serious Adverse Events (participants affected / at risk) | 28/218 | 33/218
Other Adverse Events (participants affected / at risk) | 180/218 | 178/218
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vitamin D (N=218) | Placebo: Oil (N=218)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 | 5
Vascular disorders (Vascular disorders) | 0 | 1
Surgical and medical procedures (Surgical and medical procedures) | 6 | 6
General disorders and administration site conditions (General disorders) | 1 | 3
Reproductive system and breast disorders (Reproductive system and breast disorders) | 1 | 1
Respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Psychiatric disorders (Psychiatric disorders) | 0 | 1
Cardiac disorders (Cardiac disorders) | 4 | 2
Nervous system disorders (Nervous system disorders) | 1 | 0
Ear and labyrinth disorders (Ear and labyrinth disorders) | 1 | 0
Eye disorders (Eye disorders) | 1 | 0
Gastrointestinal disorders (Gastrointestinal disorders) | 3 | 5
Hepatobiliary disorders (Hepatobiliary disorders) | 2 | 1
Skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 1 | 2
Renal and urinary disorders (Renal and urinary disorders) | 3 | 2
Endocrine disorders (Endocrine disorders) | 2 | 0
Musculoskeletal and connective tissue disorders (Musculoskeletal and connective tissue disorders) | 4 | 4
Infections and infestations (Infections and infestations) | 3 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vitamin D (N=218) | Placebo: Oil (N=218)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 18 | 11
Vascular disorders (Vascular disorders) | 2 | 1
Surgical and medical procedures (Surgical and medical procedures) | 14 | 16
Pregnancy, puerperium and perinatal conditions (Pregnancy, puerperium and perinatal conditions) | 0 | 1
General disorders and administration site conditions (General disorders) | 36 | 32
Reproductive system and breast disorders (Reproductive system and breast disorders) | 6 | 6
Respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 29 | 46
Psychiatric disorders (Psychiatric disorders) | 1 | 2
Product issues (Product Issues) | 42 | 1
Cardiac disorders (Cardiac disorders) | 9 | 7
Nervous system disorders (Nervous system disorders) | 15 | 7
Blood and lymphatic system disorders (Blood and lymphatic system disorders) | 8 | 3
Ear and labyrinth disorders (Ear and labyrinth disorders) | 7 | 4
Eye disorders (Eye disorders) | 9 | 5
Gastrointestinal disorders (Gastrointestinal disorders) | 36 | 38
Hepatobiliary disorders (Hepatobiliary disorders) | 5 | 2
Skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 35 | 22
Renal and urinary disorders (Renal and urinary disorders) | 17 | 13
Endocrine disorders (Endocrine disorders) | 44 | 99
Musculoskeletal and connective tissue disorders (Musculoskeletal and connective tissue disorders) | 39 | 37
Infections and infestations (Infections and infestations) | 57 | 55
Metabolism and nutrition disorders (Metabolism and nutrition disorders) | 2 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-01-05): https://cdn.clinicaltrials.gov/large-docs/48/NCT01748448/Prot_SAP_000.pdf